CLINICAL TRIAL: NCT00782574
Title: A Phase I Open Label, Multi Centre Study of AZD2281 Administered Orally in Combination With Cisplatin, to Assess the Safety and Tolerability in Patients With Advanced Solid Tumours
Brief Title: Phase I AZD2281/Cisplatin in Advanced Solid Tumour Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00021; 2008-000062-24 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumours; Poly(ADP ribose) polymerases; homologous deficiency; BRCA1
MeSH Terms: interventions — olaparib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Olaparib is available as a film-coated tablet containing 150 mg or 100 mg of olaparib. Subjects will be administered study treatment orally at a dose recommended by Investigator.
  Full dose: 300 mg twice daily (bid) or Reduced doses: 200 mg twice daily (bid) or 100 mg twice daily (bid).
  The planned dose of 300 mg bid will be made up of two x 150 mg tablets twice daily, with 100 mg tablets used to manage dose reductions.
  Interventions: Drug: AZD2281; Drug: Cisplatin

INTERVENTIONS:
Drug: AZD2281 — Tablets Oral BID
  Other Names: Olaparib; Lynparza
Drug: Cisplatin — IV every 3 weeks

SUMMARY:
A Phase I study to assess the safety and tolerability of AZD2281 in combination with Cisplatin in patients with advanced Solid Tumours. This is an open label-dose finding; to establish the maximum tolerated dose of AZD2281 combined with Cisplatin in patients with advanced solid tumours. Approximately 50 (max 60) patients from 2 countries will be enrolled

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Histologically confirmed metastatic cancer, not amenable to surgery or radiation therapy with curative intent
* Patients with measurable or non measurable disease according to RECIST

Exclusion Criteria:

* Less than 28 days from active therapy (ie any treatment used to treat the disease) or high dose radiotherapy
* Brain Metastases or spinal cord compression unless irradiated at least 4 weeks before entry and stable without steroid treatment for >1 week
* Persistent CTCAE Grade 2 or greater toxicities (excluding alopecia) caused by prior therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-11-12 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of AZD2281 in combination with Cisplatin (eg Adverse Events, Pharmacokinetic for AZD2281, overall response rate) to patients with advanced solid tumours. | Weekly visits for routine monitoring visits

SECONDARY OUTCOMES:
To compare exposure to AZD2281 when given alone and in combination with Cisplatin (Only in patients receiving continuous dosing of AZD2281). | PK samples taken at visit 2 and 3
To make a preliminary assessment of the anti-tumour activity of AZD2281 when given in combination with Cisplatin, by measuring overall objective response rate. | Assessed at screening, visit 9, and at end of every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Judy E Garber, Principal Investigator — Dana-Farber Cancer Institute; J Ballmana Gelpi, Principal Investigator — Vall d'Hebron
Locations (2):
- Research Site, Boston, Massachusetts, United States
- Research Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D0810C00021 redacted protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1674&filename=D0810C00021_revised_CSP_6_redacted_SECURED.pdf
- See also: CSR_Synopsis_D0810C00021.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1674&filename=D0810C00021.pdf